CLINICAL TRIAL: NCT02404805
Title: Drug Interaction Potential Between Dolutegravir and Simeprevir in HIV/Hepatitis C Virus (HCV) Seronegative Volunteers
Brief Title: Drug Interaction Potential Between Dolutegravir and Simeprevir in HIV/HCV Seronegative Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 15-0106; 152252 (Other Grant/Funding Number: ViiV Healthcare)
Record Dates: First submitted 2015-03-18; First posted 2015-04-01 (Estimated); Results first posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-02

CONDITIONS: HIV; Hepatitis C
Keywords: dolutegravir; simeprevir; HIV; HCV
MeSH Terms: conditions — Hepatitis C | interventions — dolutegravir; Simeprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1a (Experimental): Sequence 1,2,3: simeprevir only, then dolutegravir only, then both simeprevir and dolutegravir.
  Interventions: Drug: dolutegravir; Drug: simeprevir
- Sequence 1b (Experimental): Sequence 1,3,2: simeprevir only, then both simeprevir and dolutegravir, then dolutegravir only.
  Interventions: Drug: dolutegravir; Drug: simeprevir
- Sequence 2a (Experimental): Sequence 2,1,3: dolutegravir only, then simeprevir only, then both simeprevir and dolutegravir.
  Interventions: Drug: dolutegravir; Drug: simeprevir
- Sequence 2b (Experimental): Sequence 2,3,1: dolutegravir only, then both simeprevir and dolutegravir, then simeprevir only.
  Interventions: Drug: dolutegravir; Drug: simeprevir
- Sequence 3a (Experimental): Sequence 3,1,2: both simeprevir and dolutegravir, then simeprevir only, then dolutegravir only.
  Interventions: Drug: dolutegravir; Drug: simeprevir
- Sequence 3b (Experimental): Sequence 3,2,1: Both simeprevir and dolutegravir, then dolutegravir only, then simeprevir only.
  Interventions: Drug: dolutegravir; Drug: simeprevir

INTERVENTIONS:
Drug: dolutegravir — dolutegravir tablets 50mg, once daily x 7 days.
Drug: simeprevir — simeprevir tablets 150mg, once daily x 7 days.

SUMMARY:
The investigator believes simeprevir concentrations are unchanged when administered in combination with dolutegravir relative to administration alone. The investigator believes dolutegravir concentrations are unchanged when administered in combination with simeprevir. Additionally, the investigator believes simeprevir and dolutegravir are safe when administered alone and in combination.

DETAILED DESCRIPTION:
To investigate the potential for drug interactions between simeprevir and dolutegravir, participants will receive each drug alone and the drugs in combination for 7 days. The pharmacokinetics of simeprevir and dolutegravir when given in combination vs. alone will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18-60 years
* Absence of HIV-1 and HCV antibodies at screening,
* Ability and willingness to give written informed consent before the first trial-related activity.

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Active alcohol or drug abuse that, in the opinion of the investigators, would interfere with adherence to study requirements
* Participation in any investigational drug study within 30 days prior to study entry
* Currently active or chronic gastrointestinal, cardiovascular, neurologic, psychiatric, metabolic, renal, hepatic, respiratory, inflammatory, or infectious disease or malignancy requiring pharmacologic treatment, and/or if in the opinion of the investigator, would affect study participation, safety, or integrity of results
* Use of concomitant medication, including investigational, prescription, and over-the-counter products and dietary supplements with the following exceptions: aspirin, acetaminophen, ibuprofen, hormonal oral contraceptives
* Concomitant medications other than those listed above must have been discontinued at least 14 days before study entry
* Currently active dermatitis or urticaria or diagnosis of eczema or psoriasis,
* History of significant drug allergy (i.e., anaphylaxis and/or angioedema)
* Subjects with the following laboratory abnormalities at screening as defined by the 2004 Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events ("DAIDS grading table") and in accordance with the normal ranges of the trial clinical laboratory: serum creatinine grade 1 or greater (≥ 1.1 x upper limit of laboratory normal range (ULN)); hemoglobin grade 1 or greater (≤ 10.9 g/dL); platelet count grade 1 or greater (≤ 124.999 x 109/L); absolute neutrophil count grade 1 or greater (≤ 1.3 x 109/L); aspartate aminotransferase (AST) or alanine aminotransferase (ALT) grade 1 or greater (≥ 1.25 x ULN); total bilirubin grade 1 or greater (≥ 1.1 x ULN), any other laboratory abnormality of grade 2 or above.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2016-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer J Kiser, PharmD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

REFERENCES:
- [Derived] MacBrayne CE, Castillo-Mancilla J, Burton JR Jr, MaWhinney S, Wagner CB, Micke K, Fey J, Huntley RT, Larson B, Bushman LR, Kiser JJ. Small increase in dolutegravir trough, but equivalent total dolutegravir exposure with simeprevir in HIV/HCV seronegative volunteers. J Antimicrob Chemother. 2018 Jan 1;73(1):156-159. doi: 10.1093/jac/dkx344. PMID 29029135

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sequence 1a | Sequence 1b | Sequence 2a | Sequence 2b | Sequence 3a | Sequence 3b
Started | 5 | 3 | 5 | 5 | 3 | 4
Completed | 4 | 3 | 5 | 5 | 3 | 4
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1a | Sequence 1b | Sequence 2a | Sequence 2b | Sequence 3a | Sequence 3b | Total
Number analyzed (Participants) | 5 | 3 | 5 | 5 | 3 | 4 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 5 | 5 | 3 | 4 | 25
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 30.8 [18 to 60] | 34.3 [24 to 42] | 36.4 [29 to 52] | 35.6 [22 to 49] | 35.7 [26 to 45] | 33.8 [25 to 44] | 34.3 [18 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 3 | 2 | 2 | 16
  Male | 2 | 0 | 2 | 2 | 1 | 2 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ETHNICITY: CAUCASIAN | 5 | 3 | 4 | 4 | 2 | 4 | 22
  ETHNICITY: HISPANIC | 0 | 0 | 1 | 1 | 1 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 5 | 5 | 3 | 4 | 25

OUTCOME MEASURES:

1. Primary Outcome: Simeprevir AUC Pharmacokinetics
Description: Determine simeprevir area-under-the concentration time curve (AUC) when administered alone and when being co-administered with Dolutegravier.
Time Frame: Pre-dose and, 1, 2, 3, 4, 5, 6, 8, 10, 12 and 24 hours post-dose on day 7
Population: Only arms that included Simeprevir administration are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Simeprevir Administered Alone: simeprevir: simeprevir tablets 150mg, once daily x 7 days.
- Simeprevir and Dolutegravier Co-administered: Dolutegravir and simeprevir together:
  dolutegravir tablets 50mg, once daily and simeprevir tablets 150mg, once daily x 7 days.
Arm/Group | Simeprevir Administered Alone | Simeprevir and Dolutegravier Co-administered
Number analyzed (Participants) | 24 | 24
ng*h/mL | 30946 (80) | 30333 (82)

2. Primary Outcome: Dolutegravir AUC Pharmacokinetics
Description: Determine Dolutegravir area-under-the concentration time curve (AUC) when administered alone and when co-administered with simeprevir.
Time Frame: Pre-dose and, 1, 2, 3, 4, 5, 6, 8, 10, 12 and 24 hours post-dose on day 7
Population: Only arms that included Dolutegravir administration are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Dolutegravir Administered Alone: dolutegravir: dolutegravir tablets 50mg, once daily x 7 days.
- Simeprevir and Dolutegravier Co-administered: Dolutegravir and simeprevir co-administered:
  dolutegravir tablets 50mg, once daily and simeprevir tablets 150mg, once daily x 7 da
Arm/Group | Dolutegravir Administered Alone | Simeprevir and Dolutegravier Co-administered
Number analyzed (Participants) | 24 | 24
ng*h/mL | 68186 (30) | 78433 (24)

ADVERSE EVENTS:
Time Frame: Time of consenting to study exit (Phone follow up 7 days after final intensive PK visit, max 3 months)
Description: AEs were graded per the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.0, November, 2014. Available: http://rsc.tech-res.com/safetyandpharmacovigilance/.
Groups:
- Simeprevir Only: Simeprevir tablets 150mg, once daily x 7 days.
- Dolutegravir Only: Dolutegravir tablets 50mg, once daily x 7 days.
- Dolutegravir and Simeprevir Co-administered:: Dolutegravir and simeprevir co-administered:
  dolutegravir tablets 50mg, once daily, and simeprevir tablets 150mg, once daily, x 7 days
Arm/Group | Simeprevir Only | Dolutegravir Only | Dolutegravir and Simeprevir Co-administered:
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 4/25 | 7/24 | 10/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simeprevir Only (N=25) | Dolutegravir Only (N=24) | Dolutegravir and Simeprevir Co-administered: (N=24)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 3 (3)
Gastrointestinal issues (stomach pain, gas, vomiting, nausea, diarrhea) (Gastrointestinal disorders) | 2 (2) | 4 (4) | 3 (3)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Abnormal Labs (General disorders) | 1 (1) | 5 (7) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No